CLINICAL TRIAL: NCT00585078
Title: Capecitabine and Oxaliplatin in Patients With Advanced or Metastatic Pancreatic Adenocarcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Principal Investigator, Rebecca Miksad, MD, MPH, Assistant Professor, Harvard University; Attending Physician, Beth Israel Deaconess Medical Center, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 03-398; OX-03-033 (Other: sponsor)
Record Dates: First submitted 2007-12-24; First posted 2008-01-03 (Estimated); Results first posted 2017-04-10 (Actual); Last update posted 2017-04-10 (Actual); Status verified 2017-02

CONDITIONS: Pancreatic Cancer
Keywords: capecitabine; oxaliplatin
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Capecitabine; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CAPOX (Experimental): Participants self-administered capecitabine 1,000 mg/m2 orally twice daily (total daily dose 2,000 mg/m2), days 1-14 in 21-day cycles. Only 500 mg tablets were used, and doses were rounded to the nearest dose that could be administered with 500 mg tablets. Oxaliplatin 130 mg/m2 was administered intravenously on day 1 every 21 (±2) days. Treatment continued until tumor progression or toxicity requiring discontinuation of therapy.
  Interventions: Drug: Capecitabine; Drug: Oxaliplatin

INTERVENTIONS:
Drug: Capecitabine
  Other Names: Xeloda
Drug: Oxaliplatin
  Other Names: Eloxatin

SUMMARY:
There are limited treatment options available for patients with advanced pancreatic ductal adenocarcinoma (PDAC). The purpose of this study is to determine the effectiveness and safety of the drugs capecitabine and oxaliplatin in patients who have been diagnosed with advanced and metastatic PDAC treated in the first and second lines.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the response rate to capecitabine and oxaliplatin in patients with locally advanced or metastatic pancreatic adenocarcinoma Secondary
* To determine safety
* To determine overall survival
* To determine time to progression

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* At most one prior chemotherapy regimen for unresectable or metastatic disease. Any adjuvant chemotherapy must have been completed more than 12 months prior to beginning protocol therapy
* Histologically or cytologically confirmed adenocarcinoma of the pancreas
* At least one measurable lesion according to RECIST criteria that has not been irradiated
* Adequate laboratory parameters as outlined in protocol
* Anticoagulation with coumadin is permitted, but PT/INR must be monitored closely, given the drug-drug interaction between coumadin and capecitabine
* Negative serum pregnancy test within 14 days prior to registration

Exclusion Criteria:

* Pregnant or lactating women
* Life expectancy < 3 months
* Serious, uncontrolled, concurrent infection(s)
* Any prior oxaliplatin or fluoropyrimidine therapy
* More than one prior chemotherapy regimen for unresectable or metastatic disease
* Prior unanticipated severe reaction to fluoropyrimidine therapy, or known sensitivity to 5-fluorouracil or platinum compounds
* Any active second malignancy
* Clinically significant cardiac disease or myocardial infarction within the last 12 months
* Evidence of CNS metastases or history of uncontrolled seizures, central nervous system disorders or psychiatric disability
* Other serious uncontrolled medical conditions
* Major surgery within 4 weeks of the start of study treatment, without complete recovery
* Lack of physical integrity of the upper gastrointestinal tract or malabsorption syndrome
* Known, existing uncontrolled coagulopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2004-05 (Actual); Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Miksad, MD, MPH, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from May 2004 to March 2010.
Period: Overall Study
Arm/Group | CAPOX
Started | 40
Treated | 37
Toxicity Evaluable (Participants who received treatment and with toxicity data reported were evaluable for toxicity.) | 36
Response Evaluable (Per protocol, participants must have completed 2 cycles of treatment to be evaluable for response.) | 24
Completed (Since treatment was not of fixed duration, all participants were considered as 'Not Completed'.) | 0
Not Completed | 40
Not completed — Withdrawal by Subject | 4
Not completed — Poor performance status | 1
Not completed — Disease Progression | 24
Not completed — Adverse Event | 10
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Population: The analysis dataset is comprised of enrolled patients.
Arm/Group | CAPOX
Number analyzed (Participants) | 40
Age, Continuous [Median (Full Range); unit: years] | 61 [40 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 19
Region of Enrollment [Number; unit: participants]
  United States | 40
Stage [Count of Participants; unit: Participants]
  Locally Advanced | 2
  Metastatic | 38

OUTCOME MEASURES:

1. Primary Outcome: Response Rate
Description: Response rate (RR) is defined as the proportion of participants achieving partial response (PR) or complete response (CR) based on RECIST 1.0 criteria on treatment. Per RECIST 1.0 for target lesions, CR is complete disappearance of all target lesions and PR is at least a 30% decrease in the sum of longest diameter (LD) of target lesions, taking as reference baseline sum LD. To be assigned a status of CR or PR, changes in tumor measurements must be confirmed by repeat assessments performed no fewer than 4 weeks after the response criteria are first met. PR or better overall response assumes at a minimum incomplete response/stable disease (SD) for the evaluation of non-target lesions and absence of new lesions.
Time Frame: Response was assessed by computed tomography (CT) or magnetic resonance imaging (MRI) every two cycles (42 days ±2 days) on treatment. Participants received a median (range) of 2 cycles (1-12) of CAPOX.
Population: The analysis dataset is comprised of response evaluable participants which required completion of two cycles of treatment.
Measure: Number (80% Confidence Interval); unit: proportion of participants
Arm/Group | CAPOX
Number analyzed (Participants) | 24
proportion of participants | .125 [.035 to .201]

2. Secondary Outcome: Best Response
Description: Best response on treatment was based on RECIST 1.0 criteria: Complete Response (CR) is complete disappearance of all target lesions; Partial Response (PR) is at least a 30% decrease in the sum of longest diameter (LD) of target lesions, taking as reference baseline sum LD. Both require confirmation no fewer than 4 weeks apart. CR/PR assumes at a minimum incomplete response/stable disease (SD) for the evaluation of non-target lesions and absence of new lesions. Progressive disease (PD) is at least a 20% increase in the sum of longest diameter of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. PD for the evaluation of non-target lesions is the appearance of one or more new lesions and/or unequivocal progression of non-target lesions. Stable disease is defined as any condition not meeting above criteria.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | CAPOX
Number analyzed (Participants) | 24
participants
  Complete Response | 0
  Partial Response | 3
  Stable Disease | 13
  Progressive Disease | 8

3. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the time from study entry to death or date last known alive and estimated using Kaplan-Meier (KM) methods.
Time Frame: Participants were followed long-term for survival every 3 months from the end of treatment until death or lost to follow-up. Median survival follow-up was 10.8 months (95% CI: 7.1-37.7) in this study cohort.
Population: The analysis dataset is comprised of treated participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | CAPOX
Number analyzed (Participants) | 37
months | 7.4 [4.8 to 12.2]

4. Secondary Outcome: Progression-Free Survival
Description: Progression-free survival based on the Kaplan-Meier method is defined as the duration of time from study entry to documented disease progression (PD) requiring removal from treatment or death. Per RECIST 1.0 criteria: progressive disease (PD) is at least a 20% increase in the sum of longest diameter (LD) of target lesions taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. PD for the evaluation of non-target lesions is the appearance of one or more new lesions and/or unequivocal progression of non-target lesions.
Time Frame: Disease evaluations occurred every two cycles (42 days ±2 days) on treatment. In this study cohort, participants were followed for progression up to 38 months.
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | CAPOX
Number analyzed (Participants) | 24
months | 3.8 [1.3 to 6.2]

ADVERSE EVENTS:
Time Frame: Assessed each cycle on day 1 and mid-cycle (between days 10 and 14) from time of first dose and up to day 30 post-treatment. Participants received a median (range) of 2 cycles (1-12) of CAPOX.
Description: Maximum grade toxicity by type was first calculated including only adverse events with treatment-attribution of possibly, probably or definitely related to CAPOX. Serious and Other AEs were defined as grades 3-5 and grades 1-2, respectively, per CTCAEv3.The analysis dataset is comprised of all participants who started CAPOX and reported any toxicity data (toxicity evaluable). One participant was missing toxicity data.
Arm/Group | CAPOX
All-Cause Mortality (participants affected / at risk) | 0/40
Serious Adverse Events (participants affected / at risk) | 18/36
Other Adverse Events (participants affected / at risk) | 34/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CAPOX (N=36)
Hemoglobin (Blood and lymphatic system disorders) | 3
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 5
Nausea (Gastrointestinal disorders) | 6
Vomiting (Gastrointestinal disorders) | 4
Abdomen, pain (Gastrointestinal disorders) | 3
Fatigue (General disorders) | 7
Weight loss (Investigations) | 1
Metabolic/Laboratory-other (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 1
Hyperkalemia (Metabolism and nutrition disorders) | 1
Nonneuropathic generalized weakness (Musculoskeletal and connective tissue disorders) | 1
Neuropathy-sensory (Nervous system disorders) | 1
Confusion (Psychiatric disorders) | 1
Hand-foot reaction (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CAPOX (N=36)
Hemoglobin (Blood and lymphatic system disorders) | 11
Hematologic-other (Blood and lymphatic system disorders) | 2
Cardiac-other (Cardiac disorders) | 1
Hearing-other (Ear and labyrinth disorders) | 1
Vision-blurred (Eye disorders) | 1
Tearing (Eye disorders) | 2
Ocular-other (Eye disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 7
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 8
Dry mouth (Gastrointestinal disorders) | 3
Esophagitis (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 1
Muco/stomatitis (symptom) oral cavity (Gastrointestinal disorders) | 5
Nausea (Gastrointestinal disorders) | 19
Salivary (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 15
GI-other (Gastrointestinal disorders) | 9
Abdomen, pain (Gastrointestinal disorders) | 4
Fatigue (General disorders) | 19
Fever w/o neutropenia (General disorders) | 2
Rigors/chills (General disorders) | 1
Constitutional, other (General disorders) | 1
Pain-other (General disorders) | 7
Infection-other (Infections and infestations) | 2
Leukocytes (Investigations) | 5
Lymphopenia (Investigations) | 1
Neutrophils (Investigations) | 3
Platelets (Investigations) | 7
Weight loss (Investigations) | 6
INR (Investigations) | 3
PTT (Investigations) | 3
Coagulation-other (Investigations) | 1
Alkaline phosphatase (Investigations) | 2
ALT, SGPT (Investigations) | 2
AST, SGOT (Investigations) | 1
Lipase (Investigations) | 1
Metabolic/Laboratory-other (Investigations) | 2
Anorexia (Metabolism and nutrition disorders) | 15
Dehydration (Metabolism and nutrition disorders) | 5
Hypoalbuminemia (Metabolism and nutrition disorders) | 2
Hyperglycemia (Metabolism and nutrition disorders) | 4
Hypomagnesemia (Metabolism and nutrition disorders) | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 3
Hyponatremia (Metabolism and nutrition disorders) | 1
Nonneuropathic generalized weakness (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal/soft tissue-other (Musculoskeletal and connective tissue disorders) | 1
Taste disturbance (Nervous system disorders) | 4
Dizziness (Nervous system disorders) | 3
Neuropathy CN I smell (Nervous system disorders) | 1
Neuropathy-motor (Nervous system disorders) | 2
Neuropathy-sensory (Nervous system disorders) | 21
Tremor (Nervous system disorders) | 2
Neurologic-other (Nervous system disorders) | 2
Head/headache (Nervous system disorders) | 2
Insomnia (Psychiatric disorders) | 2
Depression (Psychiatric disorders) | 1
Incontinence urinary (Renal and urinary disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1
Hypopigmentation (Skin and subcutaneous tissue disorders) | 1
Nail changes (Skin and subcutaneous tissue disorders) | 1
Pruritus/itching (Skin and subcutaneous tissue disorders) | 1
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1
Hand-foot reaction (Skin and subcutaneous tissue disorders) | 8
Skin-other (Skin and subcutaneous tissue disorders) | 1
Hot flashes (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No